CLINICAL TRIAL: NCT06978296
Title: HIghly MetAstatic Life Prolonging Therapy-Resistant Prostate Cancer: Role of Stereotactic Radiotherapy for Bone and Lymph Node Metastases
Brief Title: HIghly MetAstatic Life Prolonging Therapy-Resistant Prostate Cancer: Role of Stereotactic Radiotherapy for Bone and Lymph Node Metastases (HIMARS)
Acronym: HIMARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2024-22
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer Metastatic Disease; Oligometastatic Prostate Cancer (OMPC)
Keywords: Radiotherapy; Stereotaxic; oligometastatic
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a monocentric prospective level volume escalation phase I study of radiotherapy on oligometastasis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotaxic radiotherapy (Experimental): This volume escalation will be performed until MTV is reached.
  Level cohort is defined by: volume level Irradiation volume / Bone Marrow Reserve as below:
  level -1: 20% level 1 (start level): 30% level 2: 40% level 3: 50%
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — The acceptable regimens are:
  * 27 Gy / 3 fractions / 3 fractions per week
  * 35 Gy / 5 fractions / 3 fractions per week An interval of at least 24 hours should be kept between two consecutive fractions.
  Prescription must be defined on 80% isodose or higher, maximum dose up to 130% of the isodose prescription. At least 90% of the Planning Target Volume should receive the prescribed dose. A coverage of <90% of the Planning Target Volume will be considered as acceptable deviation, and coverage of <80% of the target volume as an Unacceptable Deviation. At least 90% of the Gross Tumoral Volume should receive the prescribed dose.
  Only a part of the Gross Tumoral Volume_Total could be considered for radiation, depending on the ratio with Bone Marrow Reserve. High-risk and/or symptomatic metastases will be prioritized over other metastases.
  Anatomic bone marrow reserve (BMR) will be first determined for each patient:
  BMR = Total trabecular bone - (Total trabecular bone ∩ GTV_Total)

SUMMARY:
The investigators propose redefining this concept by focusing on volume rather than the number of metastases. To achieve this, the investigators aim to determine the Maximum Tolerated Volume (MTV) of metastatic lesions treatable with SRT (Stereotaxic radiotherapy) in a phase 1 study. In this study, the investigators will recruit patients with high-volume metastatic disease in bones or lymph nodes and progressively irradiate a volume-escalated subset of the total lesions. The selection will prioritize lesions at higher risk of causing pain or complications, such as fractures, spinal compression, or vascular compression. The investigators hypothesis is that SRT targeting multiple metastases (with a total volume ≤ MTV) will extend the duration without refractory pain and/or tumor-related complications in patients with castration-resistant and chemo-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic prostate cancer with clinical progression after the use of androgen-receptor pathway inhibitor, chemotherapy or any other life-prolonging therapy. Patient could have been treated previously by RadioLigand Therapy (RLT).
* Performance Status < 3
* Bone and/or lymph node metastases based on conventional (CT and bone scan) or metabolic imaging
* Bone and/or lymph node metastases suitable for SRT, according to the investigator
* Adequate organ function:

  1. Absolute Neutrophil Count (ANC) ≥ 1000/mm3 or
  2. Platelet Count ≥ 50 000/mm3 or
  3. Haemoglobin ≥ 8 g/dL (allowing transfusion or other intervention to achieve this minimum haemoglobin)
* Age ≥ 18 years at time of study entry
* Written informed consent obtained from the patient prior to performing any protocol-related
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patient has valid health insurance
* Life time expected > 3 months

Exclusion Criteria:

* Evidence of symptomatic metastases to the lungs, brain, peritoneum or liver
* Evidence of diffuse metastatic spread to the bone marrow (e.g. positive super bone scan) or the cerebral spinal fluid as per bone scan (no lumbar puncture required).
* Evidence of presence of symptomatic spinal cord compression with indication of neurosurgical decompression.
* Patient with symptomatic and/or high-risk tumor volume-to-bone marrow reserve ratio > 50%
* Concurrent enrolment in another clinical study, unless it is a non-therapeutic clinical study
* Mental impairment (psychiatric illness/social situations) that may compromise the ability of the patient to give informed consent and comply with the requirements of the study;
* Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship;
* Patients unable to undergo medical follow-up in the study for geographical, social or psychological reasons.
* History of another primary malignancy except for

  1. Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of SRT and of low potential risk for recurrence
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* Uncontrolled pain that contraindicates patient positioning on the radiotherapy table according to investigator
* Patient indicated to or currently treated by cytopenic treatment as chemotherapy or RadioLigand Therapy
* Patient under concomitant treatment that may generate severe gastro-intestinal disorder or genito-urinary disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated volume (MTV) | 12 weeks
  The MTV will be defined as the highest volume that can be treated with an acute toxicity of grade < 3 (CTCAE V5.0 scale) in one third of patient and will allow us to determine the recommended phase II volume under the assumption that higher volumes are likely to be more toxic. The maximum tolerated Volume (MTV) is defined as the volume at which 2 Dose-Limiting Toxicity (DLT) were observed among 3 to 6 patients.
  DLT are considered as:
  * Death clearly related to irradiation
  * Intractable pain despite oral or intravenous opioids and/or corticosteroids (EVA > 4 and increase of 2 from EVA baseline)
  * Any new grade ≥ 3 toxicity (CTCAE V5.0 scale) compared to baseline among:
    * Anemia
    * Febrile Neutropenia
    * Hemorrhage within grade ≥3 thrombocytopenia
    * Any gastro-intestinal-related disorder
    * Any genito-urinary-related disorder
    * Pneumonitis Bone marrow reserve will be determined by CT-base automatic tool.

SECONDARY OUTCOMES:
Number of toxicity related to radiotherapy as assessed by CTCAE v5.0 | through study completion
  Acute (≤ 12 weeks) and late (>12 weeks) toxicity will be evaluated according to NCI-CTCAE v5 grading
Recommended volume for irradiation by SRT for phase-II | 12 weeks
  The Recommended Volume (RV) corresponds to the volume of the level immediately below the MTV. This Recommended Volume for irradiation by SRT will then be applied for phase 2.
Pain relief assessed by EVA scale | 6 months
  Global pain evaluation (EVA) will be measured at baseline, 1-, 3- and 6-month following SRT. Score is 0 (no pain) to 10 (maximal pain)
Time to first pejorative event among tumour-related complication (bone, neurological or vascular compression) and/or death | 2 years
  Time to first worsening event due to tumor progression (as seen on thoraco-abdomino-pelvic CT scan): including bone displacement, spinal cord or neurological compression, and vasculo-lymphatic compression will be assessed.
Number of deceased patients | 2 years
  Overall survival is defined as the time interval between the date of registration and the date of death irrespective of the cause

OTHER OUTCOMES:
To assess the functioning bone marrow reserve at baseline and after SRT | Baseline and 3 months after start of SRT
  Functioning bone marrow reserve is quantified on 99Tc-sulfur colloid SPECT-CT by automatic delineation at baseline and at 3 months after SRT (GTV_Total/functioning BMR)
To compare the anatomical and functioning assessment of the bone marrow reserve | Baseline and 3 months after start of SRT
  Comparison of the tumor volume-to-bone marrow reserve ratio: GTV_total/functioning BMR and GTV_Total/anatomic BMR

CONTACTS AND LOCATIONS:
Overall Officials: Loïg Vaugier, MD, Principal Investigator — ICO
Locations (1):
- ICO, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: Undecided